CLINICAL TRIAL: NCT02560623
Title: Minimally-Invasive Detection of Barrett's Esophagus and Barrett's Esophagus Related Dysplasia/Carcinoma by a Sponge on String Device
Brief Title: A Minimally-Invasive Sponge on a String Device for Screening for Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Exact Sciences Corporation (Industry)
Responsible Party: Principal Investigator, Prasad G. Iyer, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15-004540; NCI-2022-08390 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-004540 (Other: Mayo Clinic in Rochester); P30CA015083 (NIH)
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Barrett Esophagus
Keywords: Barrett's; esophagus; reflux; esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Adenocarcinoma Of Esophagus | interventions — Biopsy; Specimen Handling; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Phase 1: Sponge on a String 25 mm 10 pores/inch (Experimental): In phase 1 of the study, subjects will be assigned to swallow a capsule sponge device 25 mm 10 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Endoscopic Procedure; Device: Swallowable Sponge Cell Sampling Device
- Phase 1: Sponge on a String 25 mm 20 pores/inch (Experimental): In phase 1 of the study, subjects will be assigned to swallow a capsule sponge device 25 mm 20 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Endoscopic Procedure; Device: Swallowable Sponge Cell Sampling Device
- Phase 2: Cases - Barrett's Esophagus (Experimental): In phase 2 of the study, additional subjects will be assigned to swallow a capsule sponge device 25 mm 10 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Interventions: Procedure: Biopsy; Procedure: Endoscopic Procedure; Device: Swallowable Sponge Cell Sampling Device
- Phase 2: Controls - No Barrett's Esophagus (Experimental): In phase 2 of the study, additional subjects will be assigned to swallow a capsule sponge device 25 mm 10 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Interventions: Procedure: Biopsy; Procedure: Endoscopic Procedure; Device: Swallowable Sponge Cell Sampling Device

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Phase 1: Sponge on a String 25 mm 10 pores/inch; Phase 1: Sponge on a String 25 mm 20 pores/inch
Procedure: Endoscopic Procedure — Undergo endoscopy
  Other Names: Endoscopic Examination; Endoscopy
Device: Swallowable Sponge Cell Sampling Device — Undergo swallowable sponge cell sampling assessment
  Other Names: Cytosponge; Swallowable Sponge; Swallowable Sponge Device

SUMMARY:
This study is being done to collect data on the potential use of a sponge on a string device as a non-invasive tool in evaluating patients with Barrett's Esophagus compared to healthy controls.

DETAILED DESCRIPTION:
This study will be conducted in two phases: Phase 1 and Phase 2. Phase 1 will consist of determining the most optimal sponge on a string design (25 mm sponge 20 pores/inch or 25 mm sponge 10 pores/inch) chosen based on participant acceptance, tolerability, mucosal irritation and DNA yield, using a randomized factorial design pilot trial. Participants will first undergo the sponge on a string test followed by clinical endoscopy. Following completion of Phase 1 trial, the most optimal sponge on a string configuration will be chosen for Phase 2. Phase 2 will be conducted using a single size sponge with the same porosity configuration selected from Phase 1. Study procedures, testing and follow up will be the same as Phase 1.

ELIGIBILITY:
Inclusion Criteria:

Subjects with known Barrett's Esophagus (BE).

* Patients with a BE segment ≥ 1cm in maximal extent endoscopically.
* Histology showing evidence of intestinal metaplasia with or without presence of dysplasia.
* Undergoing clinically indicated endoscopy. Subjects without known evidence of BE - Undergoing clinically indicated diagnostic endoscopy

Exclusion Criteria:

* Subjects with known BE.

  * Patients with prior history of ablation (photodynamic therapy, radiofrequency ablation, cryotherapy, argon plasma coagulation). Patients with history of endoscopic mucosal resection alone will not be excluded.
  * Patients with history of esophageal resection for esophageal carcinoma. Subjects with or without known evidence of BE (on history or review of medical records).
  * Pregnant or lactating females.
  * Patients who are unable to consent.
  * Patients with current history of eosinophilic esophagitis, achalasia or uninvestigated dysphagia.
  * Patients on oral anticoagulation including Coumadin, Warfarin.
  * Patients on antiplatelet agents including Clopidogrel, unless discontinued for 3 days prior to the sponge procedure.
  * Patients on oral thrombin inhibitors including Dabigatran and oral factor X a inhibitors such as rivaroxaban, apixaban and edoxaban, unless discontinued for 3 days prior to the sponge procedure.
  * Patients with history of known varices or cirrhosis.
  * Patients with history of esophageal resection for esophageal carcinoma.
  * Patients with congenital or acquired bleeding diatheses.
  * Patients with a history of esophageal squamous dysplasia.
  * Patient has known carcinoma of the foregut (pancreatic, bile duct, ampullary, stomach, or duodenum) within 5 years prior to study enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (6):
- United States (6):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic Health System - Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Northwell Health, Manhasset, New York
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iyer PG, Slettedahl SW, Mahoney DW, Giakoumopoulos M, Olson MC, Krockenberger M, Taylor WR, Foote P, Berger C, Leggett C, Wu TT, Antpack E, Falk GW, Ginsberg GG, Abrams JA, Lightdale CJ, Ramirez F, Kahn A, Wolfsen H, Konda V, Trindade AJ, Kisiel JB. Algorithm Training and Testing for a Nonendoscopic Barrett's Esophagus Detection Test in Prospective Multicenter Cohorts. Clin Gastroenterol Hepatol. 2024 Aug;22(8):1596-1604.e4. doi: 10.1016/j.cgh.2024.03.003. Epub 2024 Mar 19. PMID 38513982
- [Derived] Iyer PG, Taylor WR, Slettedahl SW, Lansing RL, Hemminger LL, Cayer FK, Mahoney DW, Giakoumopoulos M, Allawi HT, Wu TT, Wang KK, Wolfsen HC, Antpack E, Kisiel JB. Validation of a methylated DNA marker panel for the nonendoscopic detection of Barrett's esophagus in a multisite case-control study. Gastrointest Endosc. 2021 Sep;94(3):498-505. doi: 10.1016/j.gie.2021.03.937. Epub 2021 Apr 20. PMID 33857451
- [Derived] Iyer PG, Taylor WR, Johnson ML, Lansing RL, Maixner KA, Yab TC, Simonson JA, Devens ME, Slettedahl SW, Mahoney DW, Berger CK, Foote PH, Smyrk TC, Wang KK, Wolfsen HC, Ahlquist DA. Highly Discriminant Methylated DNA Markers for the Non-endoscopic Detection of Barrett's Esophagus. Am J Gastroenterol. 2018 Aug;113(8):1156-1166. doi: 10.1038/s41395-018-0107-7. Epub 2018 Jun 12. PMID 29891853

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Sponge on a String 25 mm 10 Pores/Inch: In phase 1 of the study, subjects will be assigned to swallow a capsule sponge device 25 mm 10 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Capsule Sponge Device 25 mm 10 pores/inch: Polyurethane foam sponge compressed in a vegetable material derived capsule, attached to a string. The capsule is swallowed by the patient. The shell of the capsule dissolves in the gastric fluid releasing the foam device as a sphere which is then pulled out with the attached string, providing brushing/cytology samples of the proximal stomach and esophagus.
- Phase 1:Sponge on a String 25 mm 20 Pores/Inch: In phase 1 of the study, subjects will be assigned to swallow a capsule sponge device 25 mm 20 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Capsule Sponge Device 25 mm 20 pores/inch: Polyurethane foam sponge compressed in a vegetable material derived capsule, attached to a string. The capsule is swallowed by the patient. The shell of the capsule dissolves in the gastric fluid releasing the foam device as a sphere which is then pulled out with the attached string, providing brushing/cytology samples of the proximal stomach and esophagus.
- Phase 2: Cases - Barrett's Esophagus; Phase 2: Controls - No Barrett's Esophagus: In phase 2 of the study, additional subjects will be assigned to swallow a capsule sponge device 25 mm 10 pores/inch to collect cells and cellular material from the mucosa in the esophagus prior to scheduled for a clinically indicated upper endoscopy
  Capsule Sponge Device 25 mm 10 pores/inch: Polyurethane foam sponge compressed in a vegetable material derived capsule, attached to a string. The capsule is swallowed by the patient. The shell of the capsule dissolves in the gastric fluid releasing the foam device as a sphere which is then pulled out with the attached string, providing brushing/cytology samples of the proximal stomach and esophagus.
Period: Overall Study
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch | Phase 2: Cases - Barrett's Esophagus | Phase 2: Controls - No Barrett's Esophagus
Started | 19 | 22 | 112 | 89
Completed | 19 | 20 | 112 | 89
Not Completed | 0 | 2 | 0 | 0
Not completed — Unable to swallow sponge | 0 | 1 | 0 | 0
Not completed — Intervention prior to sponge administration | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch | Phase 2: Cases - Barrett's Esophagus | Phase 2: Controls - No Barrett's Esophagus | Total
Number analyzed (Participants) | 19 | 22 | 112 | 89 | 242
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [53 to 70] | 63.5 [56.25 to 70.25] | 65.7 [57 to 72] | 58.9 [49 to 66] | 63 [54 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 20 | 47 | 83
  Male | 14 | 11 | 92 | 42 | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 112 | 89 | 242

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Would Have This Procedure Again
Description: Number of subjects that answered yes to the self-reported question "Would you choose to have this procedure again to screen for Barrett's esophagus?"
Time Frame: Within 24 hours of the capsule sponge administration
Population: Data collected and analyzed for only Phase 1: Sponge on a String 25 mm 10 pores/inch group and Phase 1:Sponge on a String 25 mm 20 pores/inch as this outcome is specific for phase 1 of the study only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch
Number analyzed (Participants) | 19 | 20
Participants | 19 | 16

2. Primary Outcome: Tolerability of Swallowing the Sponge Device
Description: Measured using a self-reported 5-item tolerability assessment rating discomfort during the procedure on a Likert scale of 0-10; 10 representing the "worst experience" and 0 the "best experience." This scale allows a comprehensive and individual assessment of the degree of pain, choking, gagging, anxiety and overall experienced during the procedure.
Time Frame: Within 24 hours of the capsule sponge administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch
Number analyzed (Participants) | 19 | 20
units on a scale
  Pain | 1 [0 to 1.5] | 0.5 [0 to 2]
  Choking | 1 [0 to 2.5] | 2 [1 to 4.25]
  Gagging | 2 [1 to 6] | 4.5 [2 to 5.5]
  Anxiety | 0 [0 to 1] | 1 [0 to 2.5]
  Overall | 0 [0 to 1] | 1.5 [0 to 5.25]

3. Primary Outcome: Mucosal Irritation
Description: Measured using a mucosal injury score (ranging from 1=no trauma to 5=severe) was scored from video recordings of the subsequent endoscopy conducted
Time Frame: Within 24 hours of the capsule sponge administration
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch
Number analyzed (Participants) | 19 | 20
score on a scale | 2 [1 to 2] | 1 [1 to 2]

4. Primary Outcome: DNA Yield
Description: Total amount of DNA obtained from esophageal cytology specimens collected by the capsule sponge devices.
Time Frame: Within 24 hours of the capsule sponge administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: μg
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch
Number analyzed (Participants) | 19 | 20
μg | 38.0 [28.5 to 51.5] | 30.8 [26.1 to 41.8]

5. Secondary Outcome: Sensitivity of Barrett's Dysplasia Detection
Description: The sensitivity methylated DNA markers detected by the capsule sponge, in making a diagnosis of BE related dysplasia will be assessed using endoscopic surveillance biopsy histology as a gold standard.
Time Frame: Within 24 hours of the capsule sponge administration
Population: Phase 2:Controls - No Barrett's Esophagus were not analyzed for this outcome due to the outcome being specific to BE related dysplasia
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Arm/Group | Phase 2: Cases - Barrett's Esophagus | Phase 2: Controls - No Barrett's Esophagus
Number analyzed (Participants) | 112 | 0
percentage of sensitivity | 92 [85 to 96] |

6. Secondary Outcome: Specificity of Barrett's Dysplasia Detection
Description: The specificity of methylated DNA markers detected by the capsule sponge, in identifying subjects without a diagnosis of BE related dysplasia will be assessed using endoscopic surveillance biopsy histology as a gold standard.
Time Frame: Within 24 hours of the capsule sponge administration
Population: Phase 2: Cases-Barrett's Esophagus were not analyzed for this outcome due to the outcome being specific to correctly identifying subjects without BE related dysplasia
Measure: Number (95% Confidence Interval); unit: percentage of specificity
Arm/Group | Phase 2: Cases - Barrett's Esophagus | Phase 2: Controls - No Barrett's Esophagus
Number analyzed (Participants) | 0 | 89
percentage of specificity |  | 94 [87 to 98]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study at approximately seven days after research procedure on all participants.
Arm/Group | Phase 1: Sponge on a String 25 mm 10 Pores/Inch | Phase 1:Sponge on a String 25 mm 20 Pores/Inch | Phase 2: Cases - Barrett's Esophagus | Phase 2: Controls - No Barrett's Esophagus
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22 | 0/112 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 5/112 | 1/89
Other Adverse Events (participants affected / at risk) | 5/19 | 8/22 | 31/112 | 30/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Sponge on a String 25 mm 10 Pores/Inch (N=19) | Phase 1:Sponge on a String 25 mm 20 Pores/Inch (N=22) | Phase 2: Cases - Barrett's Esophagus (N=112) | Phase 2: Controls - No Barrett's Esophagus (N=89)
Hospitalization after EGD/ESD procedure (Surgical and medical procedures) | 0 | 0 | 4 | 0 — Unrelated to study
Hospitalization: Distal esophageal perforation after endoscopic mucosal perforation (Surgical and medical procedures) | 0 | 0 | 1 | 0 — Unrelated to study
ER Presentation: Compliant of sore throat 3 days after procedure (Surgical and medical procedures) | 0 | 0 | 0 | 1 — Unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Sponge on a String 25 mm 10 Pores/Inch (N=19) | Phase 1:Sponge on a String 25 mm 20 Pores/Inch (N=22) | Phase 2: Cases - Barrett's Esophagus (N=112) | Phase 2: Controls - No Barrett's Esophagus (N=89)
Throat Irritation (General disorders) | 3 | 6 | 23 | 21
Pain under rib cage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Difficulty swallowing (Gastrointestinal disorders) | 1 | 0 | 3 | 3
Clearing throat (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bruise on lower lip (General disorders) | 0 | 1 | 0 | 0
Heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dark lesions distal esophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mild rectal bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Taste of blood in mouth (General disorders) | 0 | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Blood in stool (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Discomfort behind breast bone (General disorders) | 0 | 0 | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mild pain following procedure (General disorders) | 0 | 0 | 1 | 0
Slow transit time of solid food (Gastrointestinal disorders) | 0 | 0 | 1 | 0
General discomfort (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT02560623/Prot_SAP_000.pdf